Pilot Study on a Health Promotion Intervention for Ultra-Orthodox Mothers of Children With ADHD NCT06703242

Date: January 30, 2024

## Intervention protocol content outline

| Session | Objective(s) | Target behavior | Method |
|---|---|---|---|
| 1 | Create a safe emotional | Member shares thoughts and | 1) <b>Setting</b> : safe and attractive place in the school building |
| | environment to | _ | 2) Group contract: |
| | reduce<br>shame/stigma | group. | <ul><li>a) Therapist brings prepared contract which includes establishing boundaries, confidentiality, communication, norms of behavior, expectations from the group, overarching goals.</li><li>b) Members modify and agree through group discussion.</li></ul> |
| | | | 3) <b>Activity:</b> Members complete the ADHD stigma questionnaire and then have a follow up discussion |
| | | | 4) <b>Introduction to client diary:</b> A place for each member to write down their takeaways and mini goals during each session |
| 2 | Reduce ambiguity of diagnosis and behavioral | Members will use biological attribution and research-based | 1) <b>Short presentation:</b> provide background information on ADHD |
| | manifestations | descriptions/language | 2) Group Activity: |
| | | when discussing their child's ADHD | a) Analyze prepared ADHD script of behavioral manifestations |
| | | manifestations. | b) Members write a script together describing ADHD along with examples of ADHD behavioral manifestations (from personal experiences). |
| | 1 | Create a safe emotional environment to reduce shame/stigma Reduce ambiguity of diagnosis and behavioral | 1 Create a safe emotional environment to reduce group. 2 Reduce ambiguity of diagnosis and behavioral manifestations Reduce assafe thoughts and experiences to the group. Members will use biological attribution and research-based descriptions/language when discussing their child's ADHD |

| | | | 3) <b>Goal:</b> Have a real or imagined conversation with a person of their choice and describe their child's ADHD utilizing labelling/language from this session |
|---|---|---|---|
| 3 | Identify reliable resources regarding optimal and recommended | Members identify 1-2 appropriate resources for their child's ADHD challenges and/or parenting skills. | <ul><li>1) Short presentation:</li><li>a) Recommended ADHD treatment, clinical guidelines, examples of behavioral ADHD treatment options</li></ul> |
| | treatment for child's ADHD | | <ul><li>2) Reflective group activity:</li><li>a) Identify reliable sources of ADHD and health information</li></ul> |
| | Identify resources available to support mothering | | b) Recall successful past experiences finding reliable sources |
| | a child with ADHD | | <ul><li>3) Establish the group as a resource:</li><li>a) Follow up norms of communication with the group during and post intervention</li></ul> |
| | | | 4) <b>Goal:</b> each member creates an action plan to identify resource for managing their child's ADHD. |
| 4 | Modify negative beliefs about mothering and its relationship to child behavior Promote positive identity regarding | Members are able to<br>verbally de-couple<br>their child's ADHD<br>behaviors from their<br>mothering identity | 1) Group Activity: a) Members are presented with statements/depictions that reflect the cognitive bias (i.e., mothers are to blame for child's behavior) in various social contexts. b) Members generate personal examples of scenarios c) Members create alternate scenarios- role play positive reframing of belief in response to child's behavioral challenges (e.g. child is not responding to parenting |
| | their mothering role | | attempts at routinizing bedtime as opposed to self-blame 'I'm not a good enough mother to this child'- mother recognizes need for additional/knowledge/skills) |
| | | | 2) <b>Goal:</b> To notice cognitive bias(es) in their surroundings. |

| Developing strategies to manage | 5 | Understand the gap between the school's | Members will identify a person of interest in their | 1) Short presentation given along with key school staff member: Brief education about effective self-advocacy |
|---|---|---|---|---|
| child ADHD | | capabilities to meet | child's education and | 2) Role playing: |
| in the school | | their child's needs | be able to advocate for 1 of their child's | <ul><li>a) Members identify a need of their child with ADHD</li><li>b) Practice the skill of self-advocacy (multiple scenarios,</li></ul> |
| | | Increase mother | needs. | different contexts) |
| | | advocacy skills | | , |
| | | | | 3) Goal: Each member identifies in own life: |
| | | | | a) Where they want to apply this |
| Healthy | 6 | Promote | Members will | b) Create a plan 1) Short presentation: |
| mother-<br>healthy<br>child:<br>Legitimacy | O . | engagement in health promoting activities in response to their | increase engagement<br>in 1 health promoting<br>activity (subjectively<br>or objectively) | a) The parenting occupations and purposes framework b) Knowledge on link between healthy lifestyle behaviors and health outcomes |
| and importance of self-care | | caregiver role | • • | 2) <b>Group activity:</b> Adapted Occupational Questionnaire to build awareness of personal profile regarding engagement in health promoting activities and discussion |
| | | | | 3) Goal: |
| | | | | a) Each member chooses a goal* to promote their |
| | | | | engagement in a health promoting activity b) A stion plant setting + visualize implementation |
| | | | | b) Action plan: setting + visualize implementation, identify barriers, identify resources |
| | | cunations and purposes | | *Therapist provides a bank of goals to choose from. |

Notes. The parenting occupations and purposes framework (Lim et al., 2021)